CLINICAL TRIAL: NCT03270956
Title: A Phase II, Open-Label Safety and Tolerability Study of an Renal Autologous Cell Therapy (REACT) in Patients With Type 2 Diabetes and Chronic Kidney Disease (REGEN-003)
Brief Title: A Study of Autologous Renal Autologous Cell Therapy (REACT) in Patients With Diabetic Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prokidney (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REGEN-003
Record Dates: First submitted 2017-08-25; First posted 2017-09-01 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Masking Description: Open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Renal Autologous Cell Therapy (REACT) (Experimental): Renal Autologous Cell Therapy (REACT) Treatment - Patients will receive their first treatment of 2 injections of REACT as soon as REACT product is made available.
  Interventions: Biological: Renal Autologous Cell Therapy (REACT)

INTERVENTIONS:
Biological: Renal Autologous Cell Therapy (REACT) — Autologous selected renal cells (SRC)

SUMMARY:
The purpose of the present study is to assess the safety and efficacy of up to 2 injections of REACT given 6 months (+4 weeks) apart (maximum).

DETAILED DESCRIPTION:
All subjects enrolled will receive REACT. Subjects will receive their first REACT injection as soon as the REACT product is manufactured and shipped to the clinical site. After 6 months (+4 weeks), a second injection will be given, as appropriate. Each subject's baseline rate of renal decline, based on adequate historical clinical data obtained 24 months prior to screening visit, will serve as a comparator for monitoring the rate of progression of renal insufficiency over time.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female, 30 to 65 years of age on the date of informed consent.
2. The subject has an established diagnosis of T2DM.
3. The subject has an established diagnosis of diabetic nephropathy as the underlying cause of renal disease.
4. The subject has an established diagnosis of CKD not requiring renal dialysis, defined as having an eGFR between 14 and 20 mL/min/1.73m² inclusive at the Screening Visit and prior to REACT injection.
5. The subject has blood pressure less than 150/90 at the Screening Visit, prior to renal biopsy, and prior to REACT injection(s). Note BP should not be significantly below the previously recorded stable pressure.
6. A minimum of 3 measurements of eGFR or sCr should be obtained at least 3 months apart prior to the Screening Visit or within the previous 24 months to define the rate of progression of CKD. The subject should have adequate, historical clinical data to provide a reasonable estimate of the rate of progression of CKD. The Medical Monitor may be consulted to ensure there is sufficient data.

Exclusion Criteria:

1. The subject has a history of type 1 diabetes mellitus.
2. The subject has a history of renal transplantation.
3. The subject has a serum HbA1c level greater than 10% at the Screening Visit.
4. The subject has uncontrolled diabetes (defined as metabolically unstable by the Investigator).
5. The subject has hemoglobin levels less than 9 g/dL prior to each REACT injection.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Johns, Study Director — Prokidney
Locations (4):
- United States (4):
  - University of Arizona [WITHDRAWN], Tucson, Arizona
  - Boise Kidney & Hypertension Institute, Boise, Idaho
  - University of North Carolina- Chapel Hill, Chapel Hill, North Carolina
  - Vanderbilt University [WITHDRAWN], Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Renal Autologous Cell Therapy (REACT)
Started | 10
Completed | 3
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Renal Autologous Cell Therapy (REACT)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (5.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
BMI (kg/m^2) at Screening, [Mean (Standard Deviation); unit: kg/m^2] | 35.20 (8.415)
Volume (cm^3) - Treated kidney [Mean (Standard Deviation); unit: cm^3] | 180.97 (76.077)
Volume (cm^3) - Untreated kidney [Mean (Standard Deviation); unit: cm^3] | 163.93 (35.279)

OUTCOME MEASURES:

1. Primary Outcome: Procedure and/or Product Related Adverse Events
Description: Percentage of subjects with procedures and/or product related adverse events by System Organ Class and Preferred Term
Time Frame: Through 24 months following last REACT injection
Measure: Number; unit: percent of participants
Arm/Group | Renal Autologous Cell Therapy (REACT)
Number analyzed (Participants) | 10
percent of participants
  All Body Systems | 70.0
  Renal and urinary disorders | 60.0
  renal haematoma | 30.0
  subcapsular renal hematoma | 20.0
  haematuria | 10.0
  perinephric collection | 10.0
  Blood and lymphatic system disorder | 10.0
  anaemia | 10.0
  General disorders and administration site conditions | 10.0
  fatigue | 10.0
  Injury, poisoning, and procedural complications | 10.0
  procedural pain | 10.0

2. Secondary Outcome: Renal Specific Adverse Events
Description: Percentage of subjects with renal-specific adverse events by System Order Class and Preferred Term
Time Frame: Through 24 months following last REACT injection
Measure: Number; unit: percent of participants
Arm/Group | Renal Autologous Cell Therapy (REACT)
Number analyzed (Participants) | 10
percent of participants
  Renal and urinary disorders | 90.0
  End Stage Renal Disease | 50.0
  Renal haematoma | 40.0
  Acute Kidney Disease | 30.0
  Chronic Kidney Disease | 20.0
  Subcapsular renal haematoma | 20.0
  Haematuria | 10.0
  Hydronephrosis | 10.0
  perinephric collection | 10.0

ADVERSE EVENTS:
Time Frame: the day of biopsy through 24 months after the final injection of REACT, approximately 33 months
Description: All AEs that occur from the biopsy procedure, during treatment, or within 24 months following the final REACT injection, whether or not they are related to study procedures or the investigational product, must be recorded in the subject's medical records as well as the CRF provided by the Sponsor or its designee.
Arm/Group | Renal Autologous Cell Therapy (REACT)
All-Cause Mortality (participants affected / at risk) | 2/10
Serious Adverse Events (participants affected / at risk) | 8/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Autologous Cell Therapy (REACT) (N=10)
ESRD (Renal and urinary disorders) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2)
Abdominal wall abscess (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Subcapsular renal haematoma (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Autologous Cell Therapy (REACT) (N=10)
ESRD (Renal and urinary disorders) | 5 (5)
Fatigue (General disorders) | 4 (5)
Urinary tract infection (Infections and infestations) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 4 (4)
renal haematoma (Renal and urinary disorders) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
COVID-19 (Infections and infestations) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
Pyrexia (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
60-day review period can be extended an additional 30 days if Sponsor determines publication describes potentially patentable inventions. Publication not to be delayed more than 90 days after receipt of the proposed publication.

Sponsor may not require changes to the communication except to request removal of Sponsor Confidential Information.

No publication or disclosure shall be made by PI until the earlier of publication coordinated by Sponsor or 18 months after Study completion

DOCUMENTS (2):
  • Study Protocol (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT03270956/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT03270956/SAP_001.pdf